CLINICAL TRIAL: NCT03874481
Title: The Effect of Sleep Quality on Coronary Artery Disease and In Stent Restenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Hongjian Wang, Principal Investigator, China National Center for Cardiovascular Diseases
Other Study IDs: T2018-ZX026
Record Dates: First submitted 2018-11-20; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease; In-stent Restenosis
Keywords: sleep duration; sleep quality; coronary artery disease; in stent restenosis
MeSH Terms: conditions — Coronary Artery Disease; Sleep Initiation and Maintenance Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCI: Patients who had stent
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — follow up regularly for MACE

SUMMARY:
This is a cross-sectional and follow-up study. We analysis the relationship of sleep quality on coronary artery disease(CAD) and in stent restenosis(ISR). Further, we explore the mechanism of relationship between the sleep quality and CAD/ ISR by examining the biomarkers in the pathway of sleep-CAD/ISR.

DETAILED DESCRIPTION:
Background: Coronary artery disease (CAD) is the leading cause of mortality in the world. The important treatment of CAD is Percutaneous coronary intervention(PCI). However, in-stent-restenosis(ISR) is the major issue in the PCI. The factors of ISR include gender, age, diabetes, lipid ,obesity and so on.Recently, studies showed that sleep duration and sleep quality have effect on all of factors and have relationship with coronary artery calcification. We like to explore the relationship between sleep quality and CAD/ISR.

Aims:This is a cross-sectional and follow-up study. We analysis the relationship of sleep quality on coronary artery disease(CAD) and in stent restenosis(ISR). Further, we explore the mechanism of relationship between the sleep quality and CAD/ ISR by examining the biomarkers in the pathway of sleep-CAD/ISR.

Methods: We include patients who were diagnosed as CAD by coronary arteriography. Sleep duration and quality were evaluated from sleep questionnaire. During the 6 months and 9-12months, we follow up the patients who got PCI and get information of Major Adverse Cardiovascular Events (MACE) from follow-up questionnaire. On 9-12 months after PCI, coronary arteriography were produced in PCI patients. Biomarkers were tested during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Coronary artery disease
* PCI patients in the follow-up
* written informed consent

Exclusion Criteria:

* Heart failure; renal failure; secondary hypertension;valvular heart disease ;Cancer;

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Coronary arter disease
Sampling Method: Non-Probability Sample
Enrollment: 958 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
In-stent restenosis | 9-12 months from PCI
  The rate of in stent restenosis

SECONDARY OUTCOMES:
MACE | 6months, 12months
  The rate of cardiovascular(CV) death (death due to a cardiovascular cause), myocardial infarction (MI) or Severe Recurrent Ischemia requiring Urgent coronary artery Revascularization,Hospitalization for CV, Stroke, Death, Heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Hongjian Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No